CLINICAL TRIAL: NCT02566473
Title: Improving Orthopedic Outcomes Through a National TJR Registry
Brief Title: FORCE-TJR: Improving Orthopedic Outcomes Through a National TJR Registry
Acronym: FORCE-TJR
Status: Active, not recruiting | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Ayers, Principal Investigator, University of Massachusetts, Worcester
Other Study IDs: H00008642; P50HS018910 (AHRQ)
Record Dates: First submitted 2015-08-03; First posted 2015-10-02 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis
Keywords: Patient reported outcomes; Osteoarthritis; Total joint replacement
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Aim 1. Establish a national registry of diverse patients of orthopedic surgeons representing all regions of the country and varied hospital and surgeon practice settings (e.g., urban/rural, low and high volume) to ensure that registry analyses and research reflect typical clinical practice thereby providing optimal guidance for patients, clinicians, and national healthcare policymakers. Collect pre-operative and post-operative patient reported outcomes (PROs) for pain and function.

Aim 2: Develop new and transformative comparative effectiveness tools useful to both clinical practice and healthcare policy.

Aim 3. Broadly disseminate surveillance reports for adverse events, such as implant revision, hip dislocation, knee manipulation, and identify important variation to inform quality improvement priorities.

DETAILED DESCRIPTION:
Patients scheduling elective total joint replacement surgery are eligible to participate.

The Aims of the registry are as follows:

Aim 1. Establish a national registry of diverse patients of orthopedic surgeons representing all regions of the country and varied hospital and surgeon practice settings (e.g., urban/rural, low and high volume) to ensure that registry analyses and research reflect typical clinical practice thereby providing optimal guidance for patients, clinicians, and national healthcare policymakers. Collect pre-operative and post-operative patient reported outcomes (PROs) for pain and function.

Pre-surgery data. Patients will complete a set of computer-based clinical and behavioral health questions prior to surgery. A paper option is available as well. Data collected include demographics, medical and musculoskeletal comorbidities, pain and function measures.

6 month survey. Patients will receive an invitation to complete the 6 month survey either on the computer at home or on paper. This survey includes the symptom assessment and a screening survey for complications.

12 month and subsequent annual surveys. The 6 month survey will be repeated at 12 months and annually thereafter. In addition, the patient's contact information will be updated.

Oxford Knee Scale, EQ-5D Survey and Satisfaction Questions may be added to a subset of questionnaires.

Using the data collected to date from more than 25,000 patients, the investigators have identified national norms for pre-op and post-op pain and function as well as a Risk-adjustment model for outcomes.

Aim 2: Develop new and transformative comparative effectiveness tools useful to both clinical practice and healthcare policy.

Aim 3. Broadly disseminate surveillance reports for adverse events, such as implant revision, hip dislocation, knee manipulation, and identify important variation to inform quality improvement priorities.

ELIGIBILITY:
Inclusion Criteria:

* Must be scheduled elective primary or revision arthroplasty
* Must speak/read English or Spanish

Exclusion Criteria:

* Arthroplasty is scheduled due to fracture or malignancy
* Inability to provide informed consent due to dementia or cognitive impairment
* Terminal illness with life expectancy of less than 1 year
* Emergently scheduled surgery.
* Individuals who are under 18 years of age
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women older than age 18, who schedule elective primary or revision arthroplasty (total joint replacement; hip resurfacing; uni-compartmental knee procedures
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2011-04; Primary Completion 2031-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Unadjusted and risk-adjusted patient reported pain composite score, measured by the Hip disability and Osteoarthritis Outcome Score/Knee disability and Osteoarthritis Outcome Score (HOOS/KOOS) pain score | Up to 3 months prior to elective TJR surgery
  Collection of patient reported pain composite score from the HOOS/KOOS measure
Unadjusted and risk-adjusted patient reported physical function composite score, measured by the Short Form 36 (SF 36) Physical Component sub-score | Up to 3 months prior to elective TJR surgery
  Collection of patient reported physical function composite score from the SF 36 Physical Component sub-score measure
Change in unadjusted and risk-adjusted patient reported pain composite score, measured by the HOOS/KOOS pain score | 6 months post elective TJR
  Collection of patient reported pain composite score from the HOOS/KOOS measure
Change in unadjusted and risk-adjusted patient reported physical function composite score, measured by the SF 36 Physical Component sub-score | 6 months post elective TJR
  Collection of patient reported physical function composite score from the SF 36 Physical Component sub-score measure
Change in unadjusted and risk-adjusted patient reported pain composite score, measured by the HOOS/KOOS pain score | 12 months post elective TJR
  Collection of patient reported pain composite score from the HOOS/KOOS measure
Change in unadjusted and risk-adjusted patient reported physical function composite score, measured by the SF 36 Physical Component sub-score | 12 months post elective TJR
  Collection of patient reported physical function composite score from the SF 36 Physical Component sub-score measure
Change in unadjusted and risk-adjusted patient reported pain composite score, measured by the HOOS/KOOS pain score | 24 months post elective TJR
  Collection of patient reported pain composite score from the HOOS/KOOS measure
Change in unadjusted and risk-adjusted patient reported physical function composite score, measured by the SF 36 Physical Component sub-score | 24 months post elective TJR
  Collection of patient reported physical function composite score from the SF 36 Physical Component sub-score measure
Change in unadjusted and risk-adjusted patient reported pain composite score, measured by the HOOS/KOOS pain score | 36 months post elective TJR
  Collection of patient reported pain composite score from the HOOS/KOOS measure
Change in unadjusted and risk-adjusted patient reported physical function composite score, measured by the SF 36 Physical Component sub-score | 36 months post elective TJR
  Collection of patient reported physical function composite score from the SF 36 Physical Component sub-score measure
Change in unadjusted and risk-adjusted patient reported pain composite score, measured by the HOOS/KOOS pain score | 48 months post elective TJR
  Collection of patient reported pain composite score from the HOOS/KOOS measure
Change in unadjusted and risk-adjusted patient reported physical function composite score, measured by the SF 36 Physical Component sub-score | 48 months post elective TJR
  Collection of patient reported physical function composite score from the SF 36 Physical Component sub-score measure
Change in unadjusted and risk-adjusted patient reported pain composite score, measured by the HOOS/KOOS pain score | 60 months post elective TJR
  Collection of patient reported pain composite score from the HOOS/KOOS measure
Change in unadjusted and risk-adjusted patient reported physical function composite score, measured by the SF 36 Physical Component sub-score | 60 months post elective TJR
  Collection of patient reported physical function composite score from the SF 36 Physical Component sub-score measure
Change in unadjusted and risk-adjusted patient reported pain composite score, measured by the HOOS/KOOS pain score | 10 years post elective TJR
  Collection of patient reported pain composite score from the HOOS/KOOS measure
Change in unadjusted and risk-adjusted patient reported physical function composite score, measured by the SF 36 Physical Component sub-score | 10 years post elective TJR
  Collection of patient reported physical function composite score from the SF 36 Physical Component sub-score measure
Change in unadjusted and risk-adjusted patient reported pain composite score, measured by the HOOS/KOOS pain score | 15 years post elective TJR
  Collection of patient reported pain composite score from the HOOS/KOOS measure
Change in unadjusted and risk-adjusted patient reported physical function composite score, measured by the SF 36 Physical Component sub-score | 15 years post elective TJR
  Collection of patient reported physical function composite score from the SF 36 Physical Component sub-score measure
Change in unadjusted and risk-adjusted patient reported pain composite score, measured by the HOOS/KOOS pain score | 20 years post elective TJR
  Collection of patient reported pain composite score from the HOOS/KOOS measure
Change in unadjusted and risk-adjusted patient reported physical function composite score, measured by the SF 36 Physical Component sub-score | 20 years post elective TJR
  Collection of patient reported physical function composite score from the SF 36 Physical Component sub-score measure

SECONDARY OUTCOMES:
Surveillance reports for adverse events, such as implant revision, hip dislocation, knee manipulation and other adverse events. | 6 months post elective TJR
  Patients will complete questions regarding visits to the ER, hospital, day surgery and additional surgery

CONTACTS AND LOCATIONS:
Overall Officials: David Ayers, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Memorial Health Center; Arthritis and Total Joint Center, Worcester, Massachusetts, United States

REFERENCES:
- [Background] Ayers DC, Yousef M, Zheng H, Yang W, Franklin PD. The Prevalence and Predictors of Patient Dissatisfaction 5-years Following Primary Total Knee Arthroplasty. J Arthroplasty. 2022 Jun;37(6S):S121-S128. doi: 10.1016/j.arth.2022.02.077. Epub 2022 Feb 26. PMID 35227816
- [Background] Ayers DC, Yousef M, Zheng H, Yang W, Franklin PD. Do Patient Outcomes Vary by Patient Age Following Primary Total Hip Arthroplasty? J Arthroplasty. 2022 Jul;37(7S):S510-S516. doi: 10.1016/j.arth.2022.03.032. Epub 2022 Mar 12. PMID 35292339
- [Background] Ayers DC, Zheng H, Yang W, Yousef M. How Back Pain Affects Patient Satisfaction After Primary Total Knee Arthroplasty. J Arthroplasty. 2023 Jun;38(6S):S103-S108. doi: 10.1016/j.arth.2023.03.072. Epub 2023 Mar 30. PMID 37001625
- [Background] Ayers DC, Yousef M, Yang W, Zheng H. Age-Related Differences in Pain, Function, and Quality of Life Following Primary Total Knee Arthroplasty: Results From a FORCE-TJR (Function and Outcomes Research for Comparative Effectiveness in Total Joint Replacement) Cohort. J Arthroplasty. 2023 Jul;38(7 Suppl 2):S169-S176. doi: 10.1016/j.arth.2023.04.005. Epub 2023 Apr 29. PMID 37121490
- [Background] Ayers DC, Zheng H, Yang W, Yousef M. Gender Differences in Pain, Function, and Quality of Life Five Years Following Primary Total Knee Arthroplasty. J Arthroplasty. 2024 Aug;39(8S1):S100-S107. doi: 10.1016/j.arth.2024.04.031. Epub 2024 Apr 17. PMID 38640963
- [Background] Zheng H, Ash AS, Yang W, Liu SH, Allison J, Ayers DC. Strengthening Quality Measurement to Predict Success for Total Knee Arthroplasty: Results from a Nationally Representative Total Knee Arthroplasty Cohort. J Bone Joint Surg Am. 2024 Apr 17;106(8):708-715. doi: 10.2106/JBJS.23.00602. Epub 2024 Jan 25. PMID 38271493
- [Background] Yousef M, Zheng H, Yang W, Ayers DC. Predictive Factors of Pain and Functional Outcome 5 Years Following Total Hip Arthroplasty: A Prospective Function and Outcomes Research for Comparative Effectiveness in Total Joint Replacement Cohort Study. J Arthroplasty. 2024 Sep;39(9S1):S105-S111. doi: 10.1016/j.arth.2024.02.050. Epub 2024 Feb 25. PMID 38412901
- [Background] Ayers DC, Zheng H, Yang W, Yousef M. The Chitranjan S. Ranawat Award: Factors That Predict Outcome Five Years Following Total Knee Arthroplasty. J Arthroplasty. 2025 Jul;40(7S1):S12-S19. doi: 10.1016/j.arth.2025.03.006. Epub 2025 Mar 9. PMID 40068725
- See also: The Prevalence and Predictors of Patient Dissatisfaction 5-years Following Primary Total Knee Arthroplasty — https://pubmed.ncbi.nlm.nih.gov/35227816/
- See also: Do Patient Outcomes Vary by Patient Age Following Primary Total Hip Arthroplasty? — https://pubmed.ncbi.nlm.nih.gov/35292339/
- See also: How Back Pain Affects Patient Satisfaction After Primary Total Knee Arthroplasty — https://pubmed.ncbi.nlm.nih.gov/37001625/
- See also: Age-Related Differences in Pain, Function, and Quality of Life Following Primary Total Knee Arthroplasty: Results from a FORCE-TJR Cohort. Proceedings of the American Association of Hip and Knee Surgeons 2022 — http://pubmed.ncbi.nlm.nih.gov/37121490/
- See also: Gender Differences in Pain, Function, and Quality of Life Five Years Following Primary Total Knee Arthroplasty — http://pubmed.ncbi.nlm.nih.gov/38640963
- See also: Strengthening Quality Measurement to Predict Success for Total Knee Arthroplasty: Results from a Nationally Representative Total Knee Arthroplasty Cohort — http://pubmed.ncbi.nlm.nih.gov/38271493
- See also: Predictive Factors of Pain and Functional Outcome 5-year Following Total Hip Arthroplasty: A Prospective FORCE-TJR Cohort Study — http://pubmed.ncbi.nlm.nih.gov/38412901
- See also: . The Chitranjan S. Ranawat Award: Factors That Predict Outcome Five Years Following Total Knee Arthroplasty. J Arthroplasty — http://pubmed.ncbi.nlm.nih.gov/40068725